CLINICAL TRIAL: NCT06599957
Title: Innovative Drug Delivery Nanophotonic Platform for Implementation of Sarcoma Therapy
Acronym: DEEPLY
Status: Recruiting | Type: Observational
Sponsor: Istituto Ortopedico Rizzoli (Other)
Collaborators: Università Degli Studi del Sannio Dipartimento di Ingegneria Benevento (Unknown); IRCCS Istituto Romagnolo per lo Studio dei Tumori Dino Amadori Meldola (Unknown)
Responsible Party: Sponsor
Other Study IDs: DEEPLY; PNRR-POC-2023- 12377696 (Other Grant/Funding Number: Fondi POC PNRR)
Record Dates: First submitted 2024-09-10; First posted 2024-09-19 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Bone and Soft Tissue Tumors
Keywords: sarcomas; nanocarriers; therapy; nanophotonic
MeSH Terms: conditions — Soft Tissue Neoplasms; Sarcoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — This is a biological experimental prospective study on clinical specimens from patients undergoing surgery for soft tissue and bone sarcomas. The study is planned to obtain 15 biological samples suitable for the establishment of the aforementioned experimental models over its entire duration.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Bone and soft tissue sarcomas: Patients affected by sarcoma and undergoing surgical removal of the tumor or performing a biopsy will be enrolled. Only patients whose resection will provide sufficient tumor tissue that exceed what is necessary for pathological diagnosis characterization and banking will be enrolled.

SUMMARY:
DEEPLY aims to improve sarcoma therapy by the development of an innovative nanophotonic delivery approach to be applied in the future as an integrated local therapy for patients with inoperable tumors or with oligometastases. The major aim of the project is the development of innovative nanocarriers loaded with chemotherapeutic agents, whose delivery will be improved by the use of an optic fiber (optoporation). After the synthesis, and characterization of NPs, a prototype will be produced and preclinically validated on patient-derived biological material. This wide comprehensive methodological approach will ensure the obtainment of robust data to be faster exploited toward clinical applications.

ELIGIBILITY:
Inclusion Criteria:

* Patients eligible for the study will be male or female, with an age ranging from 0- to 85 years, undergoing surgery or biopsy for STSs or BSs including osteosarcomas.
* Included patients may have undergone or may be still in treatment with chemotherapy (also neo-adjuvant settings), targeted therapy, radiotherapy, or combination therapy.
* IRST will enroll only adult patients (age > 18 years).
* Signed informed consent from all subjects enrolled in the study. IOR patients will have to sign both the specific project Informed Consent and the IOR Biobank Informed consent.

Exclusion Criteria:

* Patients not affected by STSs or BSs will be excluded from the study, as well as patients with multiple primary tumors.

Ages: 2 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients affected by sarcoma and undergoing surgical removal of the tumor or performing a biopsy will be enrolled. Only patients whose resection will provide sufficient tumor tissue that exceed what is necessary for pathological diagnosis characterization and banking will be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-08-30 (Actual); Primary Completion 2026-08-30 (Estimated); Study Completion 2026-08-30 (Estimated)

PRIMARY OUTCOMES:
Primary Objective | 2 years
  The primary aim of the study will be to determine on primary cells or explants the efficacy of the innovative nanotechnology formulations established in the project.

SECONDARY OUTCOMES:
Secondary Objectives | 2 years
  The study will have the following secondary aims:
  I. to establish primary cultures and explants of human STSs and BSs including osteosarcomas, through different in vitro models (2D and 3D); II. to compare the efficacy of innovative NPs with standard and conventional chemotherapeutic drugs employed for the treatment of patients with sarcomas; III. to study the impact of a new delivery system on cancer cell lines, primary cultures and explants derived from fresh surgical specimen.

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - Istituto Ortopedico Rizzoli-OSOTT, Bologna, Emilia-Romagna
  - IRCCS Istituto Romagnolo per lo Studio dei Tumori Dino Amadori, Meldola, Emilia-Romagna